CLINICAL TRIAL: NCT05502614
Title: NEUROMOD UCon: Pilot Study of Dorsal Genital Nerve Stimulation for Management of Bladder Overactivity Following Spinal Cord Injury
Brief Title: Dorsal Genital Nerve Stimulation for Bladder Management After SCI
Acronym: NEUROMOD UCon
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Royal National Orthopaedic Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 276171
Record Dates: First submitted 2022-08-09; First posted 2022-08-16 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Spinal Cord Injuries; Neurogenic Bladder; Neurogenic Detrusor Overactivity; Neurogenic Bladder Dysfunction
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: Neuromodulation

INTERVENTIONS:
Device: Neuromodulation — Transcutaneous stimulation of the dorsal genital nerve using the Innocon Medical UCon device to provide on demand relief of bladder spasms
  Other Names: Dorsal Genital Nerve Stimulation

SUMMARY:
Following spinal cord injury signals between the brain and the bladder are disrupted. As a result the bladder often becomes overactive which can lead to the need for frequent trips to the toilet, regular incontinence episodes and a decreased quality-of-life. Neuromodulation is a therapy that aims to target the nerves that become overactive controlling the bladder, stopping the bladder overactivity on demand using an external (non-invasive) nerve stimulation box and sticker electrodes placed on the penis or clitoris.

This study is a pilot study that aims to investigate neuromodulation for improving symptoms of bladder overactivity when used by 10 people over eight weeks at home. We will assess whether using the device improves bladder capacity, incontinence, frequency of needing the toilet and whether there are any longer lasting changes after 8 weeks. Finally, the study will aim to find out the acceptability of using this type of therapy for participants and the acceptability of the device we are using.

Participants in this trial will participate over 13 weeks and need to visit our centre in Stanmore to have urodynamics tests in the 1st, 9th and 13th week. At home they will use a small stimulation device on a daily basis for 8 weeks to control overactivity in the bladder. Whilst at home they will record relevant outcomes in several three-day diaries and questionnaires. They will record baseline data before starting stimulation and for 4 weeks after.

ELIGIBILITY:
Inclusion Criteria:

* Spinal Cord Injury (suprasacral, AIS A-D);
* >18 years old, no upper age limit;
* SCI sustained >6 months ago;
* NDO;
* Capable of using the device at home either independently or with existing support.
* Male or female
* Willing and able to provide informed consent

Exclusion Criteria:

* recipient of intra-detrusor botulinum toxin injections within the last 6 months;
* previous surgical intervention on bladder sphincters;
* pregnancy;
* cardiac pacemaker;
* active sepsis;
* history of significant autonomic dysreflexia;
* poorly controlled epilepsy;
* patients with a cancerous tumour in the area of electrical stimulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-05-26 (Estimated)

PRIMARY OUTCOMES:
Change from baseline (week 1) in Maximum Cystometric capacity at post intervention (week 9) and follow up (week 13). | Week 1, 9 and 13
  During standard cystometry (retrograde filling of the bladder), maximum cystometric capacity will be defined as the volume emptied from the bladder after each fill.

SECONDARY OUTCOMES:
Maximum detrusor pressure | Week 1, 9 and 13
  Maximum recorded detrusor pressure during standard cystometry (retrograde filling of the bladder).
3 day bladder diary (3DBD) | Week 1, 2, 5, 9, 10 and 13
  3DBDs will be completed on clinically used bladder diaries. Participants will record voided volumes, urinary and faecal incontinence episodes and daily spasticity for 3 days. This will involve measuring the volume voided each time they urinate over the three days, using provided measuring equipment.
Incontinence Quality of Life (I-QoL) Questionnaire | Week 1, 5, 10 and 13
  Validated questionnaire to measure incontinence related quality of life. Scoring is 0 to 100 with higher scores representing greater quality of life.
EuroQol 5-Dimension 5-Level (EQ-5D-5L) Questionnaire | Week 1, 5, 10 and 13
  Validated questionnaire to measure general health. . Scoring is 0 to 100 with higher scores representing greater health
The Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) Questionnaire | Week 10
  Validated questionnaire to measure acceptability of the UCon device. Scoring is 1 to 5 with higher scores representing greater acceptance.
VAS treatment satisfaction | Week 10
  Visual analogue scale to assess treatment satisfaction. Scoring is 0 to 10 with higher scores representing greater satisfaction
Semi structured interview | Week 10
  The research team will conduct a semi-structured interview with the participant to explore further their experience of using DGNS and gain any insights into its use and effects we were unable to obtain from study outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Lynsey Duffell, PhD, Principal Investigator — University College, London
Locations (1):
- Royal National Orthopaedic Hospital, Stanmore, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doherty SP, Vanhoestenberghe A, Duffell LD, Hamid R, Knight SL. Ambulatory urodynamic monitoring assessment of dorsal genital nerve stimulation for suppression of involuntary detrusor contractions following spinal cord injury: a pilot study. Spinal Cord Ser Cases. 2020 Apr 30;6(1):30. doi: 10.1038/s41394-020-0279-4. PMID 32355163